CLINICAL TRIAL: NCT04249843
Title: A First-in-Human, Phase 1a/1b, Open Label, Dose-Escalation and Expansion Study to Investigate the Safety, Pharmacokinetics, and Antitumor Activity of the RAF Dimer Inhibitor BGB-3245 in Patients With Advanced or Refractory Tumors
Brief Title: Study of Safety, Pharmacokinetics, and Antitumor Activity of BGB-3245 in Participants With Advanced or Refractory Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated by the sponsor for reasons unrelated to safety.
Sponsor: MapKure, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BGB-3245-AU-001
Record Dates: First submitted 2020-01-21; First posted 2020-01-31 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Solid Tumor; B-Raf Mutation-Related Tumors
Keywords: BGB3245; BRAF inhibitor; BRAF; KRAS; NRAS; Mitogen Activated Protein Kinase (MAPK) Pathway; BRAF fusion; BRAF Class II

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1a: Dose Escalation (Experimental): BGB-3245 administered orally (PO)
  Interventions: Drug: BGB-3245
- Phase 1b, Group 1: Dose Expansion (Experimental): BGB-3245 administered orally (PO)
  Interventions: Drug: BGB-3245

INTERVENTIONS:
Drug: BGB-3245 — administered orally (PO)
  Other Names: Brimarafenib

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and antitumor activity of BGB-3245 in participants with advanced or refractory solid tumors

ELIGIBILITY:
Key Inclusion Criteria:

1. Participants with histologically confirmed advanced or metastatic solid tumor who had disease progression during or after systemic anticancer therapies that previously demonstrated clinical benefit (eg, improved survival) in a representative population, or are unable to receive standard therapy(ies). In addition, participants must meet the following eligibility criteria for the corresponding phase of the study:

   1. Phase 1a: participants with a known mutation status and tumor harboring an oncogenic mutation of the v-RAF murine sarcoma viral oncogene homolog B (BRAF) gene (the mutations of primary interest are the BRAF Class II mutation, Class III mutation or BRAF fusion). In addition, participants with tumors harboring the mutation of the neuroblastoma RAS viral oncogene homolog (NRAS) gene or the Kirsten rat sarcoma virus oncogene homolog (KRAS) are eligible for Part 1a. For participants with KRAS mutations, tumor types of colorectal cancer (CRC) and pancreatic cancer are excluded.
   2. Phase 1b: participants must have a known mutation status and meet one of the following criteria according to the group they are enrolled into:

   I. Group 1: participants with tumor types other than CRC that harbor BRAF V600 mutations who have been treated and progressed on prior BRAF and/or mitogen activated protein kinase (MEK) inhibition.

   II. Group 2: participants with advanced solid tumors harboring a BRAF Class II mutation or a BRAF fusion mutation.

   III. Group 2 BRAF Fusion Expansion: Participants with advanced solid tumors harboring a BRAF fusion mutation
2. Participants must provide archival tumor tissue or agree to a fresh tumor biopsy for mutation and biomarkers analysis (fresh tumor biopsies are strongly recommended)
3. Participants must have radiologically measurable disease as defined by RECIST v1.1
4. Eastern Cooperative Oncology Group (ECOG) performance status of ≤1
5. Adequate organ function and no transfusions within 14 days of first dose

Key Exclusion Criteria :

1. Participants receiving cancer therapy (chemotherapy or other systemic anticancer therapies, immunotherapy, radiation therapy, or surgery) at the time of Cycle 1 Day 1.
2. All participants who have received prior systemic anticancer treatment within the following time frames will be excluded:

   1. Systemic chemotherapy within 4 weeks or 6 weeks for nitrosourea, mitomycin prior to Cycle 1 Day 1; and
   2. Biologic therapy (i.e., antibodies), continuous or intermittent small-molecule therapies, or any other investigational agents within a period of 5 times the half-life of the agent or ≤4 weeks (whichever is shorter) prior to Cycle 1 Day 1.
3. Severe or uncontrolled systemic disease.
4. Clinically significant cardiac disease within 6 months of signing the ICF
5. CNS metastases, leptomeningeal carcinomatosis or untreated spinal cord compression.
6. Any unstable, preexisting major medical condition, including known human immunodeficiency virus (HIV) or active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
7. Systemic anti-cancer therapy within 2 weeks or 5 half-lives before first dose.
8. Major surgical procedure or significant traumatic injury within 4 weeks prior to the first dose or anticipates need for major surgery while on study.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2025-08-04 (Actual); Study Completion 2025-08-04 (Actual)

PRIMARY OUTCOMES:
Phase 1a: Number of Participants and Severity Experiencing Adverse Events (AEs) | Up to 30 days after the last dose of study drug
Phase 1a: Number of Participants and Severity Experiencing Serious Adverse Events (SAEs) | Up to 30 days after the last dose of study drug
Phase 1a: number of Participants Experiencing AEs meeting protocol defined Dose-Limiting Toxicity (DLT) criteria | From Cycle 1 Day to the end of Cycle 1 (Cycle 1 is 30 days)
Phase 1a: Maximum Tolerated Dose (MTD) of BGB-3245, and the recommended Phase 2 Dose (RP2D) for BGB-3245 | From Cycle 1 Day to the end of Cycle 1 (Cycle 1 is 30 days)
  The MTD is defined as the highest dose evaluated for which the estimated toxicity rate is closest to the target toxicity rate of 33%.
Phase 1b: Recommended Phase 2 dose (RP2D) of BGB-3245 | From Cycle 1 Day to the end of Cycle 1 (Cycle 1 is 30 days)
  The highest dose evaluated for which the estimated toxicity rate is closest to the target toxicity rate of 33%
Phase 1b: Objective Response Rate (ORR) as assessed by the investigator | Up to 24 months
  ORR is defined as the percentage of participants with partial or complete response, as assessed by the investigator
Phase 1b: Further review of the ORR | Up to 24 months
  ORR is defined as the percentage of participants with partial or complete response in up to 15 participants with tumors harboring BRAF fusion mutations

SECONDARY OUTCOMES:
Phase 1a: Overall Response Rate (ORR) as Assessed by the Investigator | Up to 24 months
Phase 1a: Duration of Response (DOR) as Assessed by the Investigator | Up to 24 months
Phase 1a: Clinical Benefit Rate (CBR) as Assessed by the Investigator | Up to 24 months
Phase 1a: Best Overall Response (BOR) as Assessed by the Investigator | Up to 24 months
Phase 1a: Duration of Stable Disease (DSD) | Up to 24 months
Phase 1a: Progression Free Survival (PFS) | Up to 24 months
Phase 1a: Plasma Concentration of BGB-3245 | Within 60 minutes predose up to 72 hours postdose
Phase 1a: Maximum Observed Plasma Concentration (Cmax) of BGB-3245 | Within 60 minutes predose up to 72 hours postdose
Phase 1a: Time to Maximum Plasma Concentration (Tmax) of BGB-3245 | 60 minutes predose up to 72 hours postdose
Phase 1a: Time Taken for Half the Initial Dose Administered To Be Eliminated From The Body (T1/2) of BGB-3245 | 60 minutes predose up to 72 hours postdose
Phase 1a: Area Under the Concentration-Time Curve of 0-infinity Days (AUC0-inf) of BGB-3245 | 60 minutes predose up to 72 hours postdose
Phase 1a:Area Under the Concentration-Time Curve of 0-Last hour (AUC0-last) of BGB-3245 | 60 minutes predose up to 72 hours postdose
Phase 1a: Drug Clearance (CL/F) of BGB-3245 | 60 minutes predose up to 72 hours postdose
Phase 1a: Apparent Volume of Distribution (Vz/F) of BGB-3245 | 60 minutes predose up to 72 hours postdose
Phase 1a: Steady State Area Under the Concentration-Time Curve of 0- Last hour (AUCLast, ss) of BGB-3245 | 60 minutes predose up to 72 hours postdose
Phase 1a: Steady State Maximum Observed Plasma Concentration (Cmax, ss) of BGB-3245 | 60 minutes predose up to 72 hours postdose
Phase 1a: Steady State Time to Maximum Plasma Concentration (Tmax, ss) of BGB-3245 | 60 minutes predose up to 72 hours postdose
Phase 1b: Progression-free survival (PFS) as Assessed by the Investigator | Up to 36 months
Phase 1b: Duration of Response (DOR) as Assessed by the Investigator | Up to 24 months
Phase 1b: Disease-Control Rate (DCR) as Assessed by the Investigator | Up to 24 months
Phase 1b: Duration of Stable Disease (DSD) as Assessed by the Investigator | Up to 24 months
Phase 1b: Clinical Benefit Rate (CBR) as Assessed by the Investigator | Up to 24 months
Phase 1b: Overall Survival | Up to 36 months
Phase 1b: Number of Participants Experiencing Adverse Events (AEs) | Up to 30 days after the last dose of study drug
Phase 1b: Number of Participants Experiencing Serious Adverse Events (SAEs) | Up to 30 days after the last dose of study drug
Phase 1b: Plasma Concentration of BGB-3245 | 60 minutes predose up to 3 hours postdose
Phase 1b: Steady State Trough Observed Plasma Concentration (Ctrough, SS) of BGB-3245 | 60 minutes predose up to 72 hours postdose

CONTACTS AND LOCATIONS:
Locations (9):
- United States (5):
  - Cedars Sinai Medical Center, Beverly Hills, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - MD Anderson, Houston, Texas
  - University of Virginia Comprehensive Cancer Centre, Charlottesville, Virginia
- Australia (4):
  - Blacktown Hospital, Blacktown, New South Wales
  - The Kinghorn Cancer Centre, St Vincent Hospital Sydney, Sydney, New South Wales
  - One Clinical Research, Nedlands, Perth
  - Peter MacCallum Cancer Centre, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: Yes